CLINICAL TRIAL: NCT04391530
Title: The Effect of Breath Therapy and Emotional Freedom Technique on Public Speaking Anxiety in Turkish Nursing Students: A Randomized Controlled Study
Brief Title: The Effect of Breath Therapy and Emotional Freedom Technique on Public Speaking Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Berna Dincer, Assistant Prof., Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 42432569
Record Dates: First submitted 2020-05-06; First posted 2020-05-18 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Public Speaking; Anxiety; Emotional Stress
Keywords: Public Speaking Anxiety; Emotional freedom technique; stress; nursing students
MeSH Terms: conditions — Speech; Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Students who meet the inclusion criteria for the research will use the Random.org website to allocate students to the breath therapy, Emotional Freedom Technique and Control group with student numbers in the class list.
Who Masked: Outcomes Assessor
Masking Description: the analysis of the research will be done by the other researcher, not by the researcher who applied it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- emotional freedom technique group (Experimental): The EFT application will be implemented by the researcher who has been trained in this subject, in the most quiet and calm environment possible, in a position where the individuals are comfortable. There are basic steps to be followed in EFT application. Thought Field Therapy (TFT), developed by Callahan, based on Craig, uses different click points for specific psychological conditions, while EFT has 12 energy click points in the same specified order to treat every emotional problem, It is called 'Basic Recipe'
  Interventions: Behavioral: emotional freedom technique, breathing therapy
- Breathin therapy group (Experimental): Breathing therapy: the basic recipe After applying pre-test forms to students, the hall will be quiet and dim. In this study, breathing exercise application will be performed in three stages as (1) relax, (2) deep breath and (3) feel yourself.
  Interventions: Behavioral: emotional freedom technique, breathing therapy
- Control group (No Intervention): No intervention was made to the students in the control group.

INTERVENTIONS:
Behavioral: emotional freedom technique, breathing therapy — emotional freedom technique, breathing therapy
  Arms: Breathin therapy group; emotional freedom technique group

SUMMARY:
Introduction Public Speaking Anxiety (PSA), also referred to as public speaking anxiety, is a costly (Lépine, 2002) and disabling fear (Blöte et al., 2009), with prevalence rates ranging from 21 (Pollard and Henderson, 1988) to 33% (Stein et al., 1996; D'El Rey and Pacini, 2005) in community samples. FoPS has been reported as the single most commonly feared situation in both university and community samples (Pollard and Henderson, 1988; Holt et al., 1992; Stein et al., 1996; Tillfors and Furmark, 2007).EFT is an energy psychotherapy derivative application consisting of cognitive and somatic components used to improve personal negative emotions and related emotional and physical ailments.It is reported that the most recognized and used EFT among Energy Therapies is an effective method especially on anxiety, depression, burnout, stress management, and fears (Feinstein 2008; Irmak Vural & Aslan, 2018; Sezgin, 2017; Sezgin & Özcan, 2009).Breatihin therapy is another one. Purpose of the study The current study aims to determine the effect of the Breath Therapy and Emotional Freedom Technique on public speaking anxiety in Turkish Nursing Students.

The purpose of the study was to evaluate two research hypotheses as follows:

H1: Emotional freedom technique is effective in reducing public speaking anxiety H2: Breath Therapy is effective in reducing public speaking anxiety A randomized controlled experimental research design will be used. The study complied with the guidelines of the Consolidated Standards of Reporting Trials (CONSORT) checklist. The data will be collected with demographic information form, Subjective Discomfort Unit Scale, The State-Trait Anxiety Inventory, and Speech Anxiety Scale.demographic information form: This form contains 5 questions including the age, gender, economic status, place of residence of students in the form developed by the researchers.

Subjective Units of Disturbance Scale SUDS. It was developed by Wolpe (1970). This scale, which is used in energy therapies and evaluates the individual's own discomfort, is scored between 0 and 10. 0 no discomfort 10 is considered to be unbearable discomfort (Wolpe, 1973). The individual should evaluate the discomfort he feels at that moment and give a score. This score serves as a concrete and basic starting point for the patient's condition at the time of application and reflects the change at the end of the application. According to the Church; EFT; Individuals' discomfort assessments are made using the Subjective Units of Disturbance (SUD) scale used by Wolpe (Church, 2013a).

he State-Trait Anxiety Inventory (STAI Tx-1 and Tx-2) It was developed by Spilberg et al to detect the state and trait anxiety levels of individuals. Its validity and reliability in Turkish was done by Öner and Lecompte. The scale consists of a total of 40 questions, 20 questions of state anxiety and 20 questions of constant anxiety. State anxiety scale; to state how the person feels at any time and under any circumstances; It is asked to answer taking into account the feeling related to the situation. On the scale of trait anxiety; one is often expected to interpret how he feels. There are positive and negative expressions on the scale. These statements; are expressed as plain and inverted expressions. Straight expressions, negative emotions; reversed statements reflect positive emotions. There are 8 reversed statements on the state anxiety scale and 7 on the trait anxiety scale. Items on the state anxiety scale 1, 2, 5, 8, 10, 11, 15, 16, 19, 20, and on the trait anxiety scale 1,6,7,10,13,16,19. items are reversed statements. The emotions, thoughts and behaviors stated in the state anxiety scale are answered as 1: none, 4: completely according to the violence level of the experiences. Feelings, thoughts and behaviors stated in the trait anxiety scale are also marked as 1-almost never, 4-almost always according to the frequency level. For both scales; 0-19 points (none), 20-39 points (mild), 40-59 points (moderate), 60- 79 points (severe), 80 points and above are considered as very severe anxiety. Cronbach alpha value of the state anxiety scale was 0.93; The Cronbach alpha value of the trait anxiety scale is 0.94 (Öner, 1998). In the present study, Cronbach's alpha value was found to be 0.81 for the STAI Tx-1 and 0.76 for the STAI Tx-2.

Speech Anxiety Scale (CUR): It was developed by Yaman and Sofu (2013) to evaluate students' speech anxiety levels. The scale consisting of 25 items is scored as 5-point Likert type and 1: strongly disagree, 4: strongly agree. In the scale, items 5, 6, 9, 10, 13 and 14 are reversed. A high score indicates that the person's anxiety to speak is high. Cronbach alpha value of the scale was found to be 0.79. In this study, Cronbach alpha value is 0.78.

DETAILED DESCRIPTION:
The criteria for inclusion in the research are a) being 18 years of age and over b) not having any psychiatric diagnosis c) not having taken a course or lesson about coping with anxiety and stress d) not speaking before the community e) volunteering to participate in the study .

Procedure The study will be carried out before the presentations on the prevention of chronic diseases within the scope of the Chronic Diseases course. 3 separate halls will be set up for the intervention and control groups to make their presentations. Students will start working after being taken to the halls set up for them.

Demographic information form, Subjective Discomfort Unit Scale (SUD), STAI-I and STAI-II and Speech Anxiety scales will be applied to the students in the EFT intervention group. Later, information about the EFT method to be used within the scope of the research will be given. One EFT session (25 minutes) was held once. After applying SUD, STAI-I and STAI-II and Speech Anxiety scales as a final test, students in the EFT group will make their speeches in front of the community.

Demographic information form, Subjective Discomfort Unit Scale (SUD), STAI-I and STAI-II and Speech Anxiety scales will be applied to the students in the breathing exercise intervention group. Later, information will be given about the breathing exercise method to be used in the research. Students will be given one breathing exercise session (25 minutes). After applying SUD, STAI-I and STAI-II and Speech Anxiety scales as the final test, students in the breathing exercise group will have their speeches in front of the community.

Demographic information form, Subjective Discomfort Unit Scale (SUD), STAI-I and STAI-II and Speech Anxiety scales were applied to the students in the control group. No intervention was made to the students in the control group. 25 minutes after the pretest application, SUD, STAI-I and STAI-II and Speech Anxiety scales were applied as posttest. Then the students in the control group made their speeches in front of the community.

EFT tapping: the basic recipe The EFT application will be implemented by the researcher who has been trained in this subject, in the most quiet and calm environment possible, in a position where the individuals are comfortable. There are basic steps to be followed in EFT application. Thought Field Therapy (TFT), developed by Callahan, based on Craig, uses different click points for specific psychological conditions, while EFT has 12 energy click points in the same specified order to treat every emotional problem, It is called 'Basic Recipe' (Craig, 2004).

While applying the Basic Recipe, the following steps are followed;

1. Determination of SUD level (Student makes the scoring of the problem he feels on the scale between zero and ten points.)
2. Installation (The general structure is "I accept myself deeply and completely despite this ……….".
3. Clicking the meridian points in order (The points given in Figure 2 are clicked.)
4. Nine Gamut procedures (Some eye movements, murmurs and counts are made while clicking on the Gamut point in hand.)
5. Clicking the meridian points in order again
6. Control of differentiation at the level of discomfort with SUD again (Craig, 2004; Church, 2004; Craig, 2017).

Implementing the batting series: With the index finger and middle finger, EFT points (Figure 2) are struck without hurt but with precise strokes. EFT points are the end points of the energy meridians. These endpoints are close to the surface of the body and are therefore more easily accessible than other buried points. Strikes at EFT points compensate for any possible disorders. At each point, the problem statement is repeated aloud (if possible).

Breathing therapy: the basic recipe After applying pre-test forms to students, the hall will be quiet and dim. In this study, breathing exercise application will be performed in three stages as (1) relax, (2) deep breath and (3) feel yourself. Relaxing music including bird sounds and water sounds will be used to ensure the concentration and focus of the participants. It will be said to breathe deeply and feel it

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. no psychiatric diagnosis
3. no history or course about coping with anxiety and stress
4. not speaking before the community
5. volunteering to participate in the study

Exclusion Criteria:

1. not wanting to speak in public
2. not volunteering to participate in the study

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-06-05 (Estimated); Primary Completion 2020-06-10 (Estimated); Study Completion 2020-11-10 (Estimated)

PRIMARY OUTCOMES:
EFT is an energy psychotherapy derivative application consisting of cognitive and somatic components used to improve personal negative emotions and related emotional and physical ailments. EFT is effective reduce Public Speaking Anxiety | two months
  Speech Anxiety Scale (SAS): A high score indicates that the person's anxiety to speak is high.
EFT is an energy psychotherapy derivative application consisting of cognitive and somatic components used to improve personal negative emotions and related emotional and physical ailments. EFT is effective reduce Subjective Units of Disturbance | two months
  Subjective Units of Disturbance Scale SUDS scored between 0 and 10. EFT; evaluations of the individual who are disturbed are made by using the subjective units of disturbance scale
EFT is an energy psychotherapy derivative application consisting of cognitive and somatic components used to improve personal negative emotions and related emotional and physical ailments. EFT is effective reduce state Anxiety | two months
  The State-Trait Anxiety Inventory (STAI Tx-1 and Tx-2): The scale consists of a total of 40 questions, 20 questions of state anxiety and 20 questions relate to constant anxiety. State anxiety scale; to state how the person feels at any time and under any circumstances
Breath Therapy, on the other hand, is a meditation that works both with the mind and respiratory organs and provides regulation of breathing. Breath Therapy is effective reduce Public Speaking Anxiety | two months
  Speech Anxiety Scale (SAS): A high score indicates that the person's anxiety to speak is high.
Breath Therapy, on the other hand, is a meditation that works both with the mind and respiratory organs and provides regulation of breathing. Breath Therapy is effective reduce subjective Units of Disturbance | two months
  Subjective Units of Disturbance Scale SUDS scored between 0 and 10. EFT; evaluations of the individual who are disturbed are made by using the subjective units of disturbance scale
Breath Therapy, on the other hand, is a meditation that works both with the mind and respiratory organs and provides regulation of breathing. Breath Therapy is effective reduce state Anxiety | two months
  The State-Trait Anxiety Inventory (STAI Tx-1 and Tx-2): The scale consists of a total of 40 questions, 20 questions of state anxiety and 20 questions relate to constant anxiety. State anxiety scale; to state how the person feels at any time and under any circumstances

IPD SHARING:
Plan to Share IPD: Undecided